CLINICAL TRIAL: NCT03050970
Title: Performance of a Minor Head Trauma Clinical Decision Rule Dedicated to Children Younger Than Two Years: A National Prospective Multicenter Study
Brief Title: Infant Minor Head Trauma Clinical Decision Rule
Acronym: PELICAN
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Francophone Pediatric Resuscitation and Emergency Group (GFRUP) (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-A00629-42; NI 15019 - AOM 15311 (Other: Assistance-Publique Hôpitaux de Paris)
Record Dates: First submitted 2017-01-31; First posted 2017-02-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Head Trauma
Keywords: minor head trauma; child; age less than 2 years; Clinically-important traumatic brain injury (ciTBI); Computed tomography scan; Radiation exposure from CT scans
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to validate a clinical decision rule for the management of minor head trauma in infants aged less than two years, constructed with the intention of minimizing the rate of computed tomography scans ordering.

DETAILED DESCRIPTION:
Apparently minor head trauma (MHT), defined by a Glasgow coma scale score (GCS) of 14-15, is the most frequently assessed group among the population of children attending Emergency Department (ED) for head trauma. Less than 1% of children with MHT have a clinically important traumatic brain injury (ciTBI) that is requiring immediate and specific care, especially neurosurgery. Those ciTBI should be identified rapidly. Assessment of children < 2 years is particularly difficult. This may promote excessive computed tomography (CT) scans ordering in this age group, while the youngest are the most sensitive to the risk of secondary malignity induced by ionizing radiation from CT scan. In USA, 31% of children < 2 years with MHT undergo CT scan. Data for CT scan use in France are unavailable and subjected to practice variations. The predictive values of TBI clinical variables such as vomiting, immediate loss of consciousness, impact seizure, severe injury mechanism, scalp hematoma or skull fracture, are controversial. A short clinical observation of children with such signs or post-traumatic symptoms before making the decision regarding CT scan ordering seems to be beneficial, allowing selective CT scan use for children whose symptoms fail to resolve. To improve patient care, clinical decision rules attempting to risk-stratify the need for a scan have emerged in the literature.

Age-based PECARN rule derived and validated in the larger cohort of 10 718 children < 2 years is the reference in the management of minor head trauma. The PECARN rule identifies ciTBIs with an optimal sensitivity but with a high rate of normal scans or identifying a non-significant lesion (expected CT scans rate: 23%; ciTBI: 0,85%). This North American rule is recommended by the Emergency Medicine French Society for the management of minor head injury. This study aims to evaluate the performance of the PELICAN rule, a decision rule for the management of apparently minor head trauma in children < 2 years that proposes targeted indications for CT scan use and defines precise indications for clinical observation. The PELICAN rule was built after a literature review of the predictive values of TBI clinical variables with the intention of minimizing the CT scans rate without missing any ciTBI.

The primary objective is to assess the performance of the PELICAN clinical prediction rule for identifying clinical-important traumatic brain injuries after apparently minor head trauma (GCS 14-15) in infants less than 2 years. The performance of the PECARN TBI prediction rule when applied to a large national French population will also be assisted and compared to that of PELICAN rule in terms of security, efficacy and expected impact on CT ordering.

ELIGIBILITY:
Inclusion Criteria:

* Child aged less than 2 years presenting to pediatric emergencies for evaluation within 24 hours of an apparently minor blunt head trauma, defined by a pediatric Glasgow coma scale score of 14 or 15 at initial clinical assessment
* Non opposition from parents to their child inclusion and collect of these data
* Child with social insurance

Exclusion Criteria:

* Trivial head injury
* Neurosurgical history
* Pre-existing neurological disorder
* Bleeding disorder
* Suspected child abuse
* Open fracture
* Penetrating skull injury
* Polytrauma and substantial non cranial serious injury
* Isolated facial trauma
* Imaging performed before ED visit
* Prior inclusion of the child in the study

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants aged less than two years attending at emergency departments
Sampling Method: Non-Probability Sample
Enrollment: 8802 (Actual)
Dates: Start 2017-02-11 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Presence of a clinically-important traumatic brain injuries (ciTBI) | 7 days after head trauma
  Clinically-important traumatic brain injury defined by: death, intubation > 24h, neurosurgical intervention and/or admission > 2 nights for head injury with traumatic brain injury on CT scan

SECONDARY OUTCOMES:
Rate of CT scans that would be recommended by the PELICAN rule applied in the study population | Initial emergency clinical evaluation
  Assessment of the number of children with any of the PELICAN predictive variables recommending CT scan ordering
Rate of CT scans that would be recommended by the PELICAN rule applied in the study population | 24 hours following the initial evaluation
  Assessment of the number of children with any of the PELICAN predictive variables recommending CT scan ordering
Number of patients with any of the six predictive variables of PECARN rule and classification in each risk-level group | Initial emergency clinical evaluation
  Performance of the age-based PECARN TBI prediction rule for identifying ciTBI
Number of patients with TBI on CT undergoing neurosurgery | 7 days after head trauma
  TBI outcomes of children < 2 years
Rate of CT scan use in practice | 7 days after head trauma
  to analyse the different management care strategies applied to a large national French observational study population
Number of patients with a non-clinically significant TBI identified on CT scan who would have been missed by the PELICAN rule | 7 days after head trauma
  Presence of a TBI on CT scan that doesn't result in death, intubation < 24h, neurosurgery and/or admission over 2 nights, in a patient who had no PELICAN predictors recommending CT scan.
  Presence in these patients of post-traumatic signs or symptoms requiring admission or any specific therapy
Rate of Admission for short ED clinical observation expected by the application of PELICAN rule | 24 hours after head trauma
  Presence of a PELICAN variable recommending short clinical observation

CONTACTS AND LOCATIONS:
Overall Officials: Gérard CHERON, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Géraldine PATTEAU, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pediatric Emergency Department - Necker-Enfants malades Hospital -, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuppermann N, Holmes JF, Dayan PS, Hoyle JD Jr, Atabaki SM, Holubkov R, Nadel FM, Monroe D, Stanley RM, Borgialli DA, Badawy MK, Schunk JE, Quayle KS, Mahajan P, Lichenstein R, Lillis KA, Tunik MG, Jacobs ES, Callahan JM, Gorelick MH, Glass TF, Lee LK, Bachman MC, Cooper A, Powell EC, Gerardi MJ, Melville KA, Muizelaar JP, Wisner DH, Zuspan SJ, Dean JM, Wootton-Gorges SL; Pediatric Emergency Care Applied Research Network (PECARN). Identification of children at very low risk of clinically-important brain injuries after head trauma: a prospective cohort study. Lancet. 2009 Oct 3;374(9696):1160-70. doi: 10.1016/S0140-6736(09)61558-0. Epub 2009 Sep 14. PMID 19758692
- [Background] Schonfeld D, Bressan S, Da Dalt L, Henien MN, Winnett JA, Nigrovic LE. Pediatric Emergency Care Applied Research Network head injury clinical prediction rules are reliable in practice. Arch Dis Child. 2014 May;99(5):427-31. doi: 10.1136/archdischild-2013-305004. Epub 2014 Jan 15. PMID 24431418
- [Background] Bressan S, Romanato S, Mion T, Zanconato S, Da Dalt L. Implementation of adapted PECARN decision rule for children with minor head injury in the pediatric emergency department. Acad Emerg Med. 2012 Jul;19(7):801-7. doi: 10.1111/j.1553-2712.2012.01384.x. Epub 2012 Jun 22. PMID 22724450
- [Background] Osmond MH, Klassen TP, Wells GA, Correll R, Jarvis A, Joubert G, Bailey B, Chauvin-Kimoff L, Pusic M, McConnell D, Nijssen-Jordan C, Silver N, Taylor B, Stiell IG; Pediatric Emergency Research Canada (PERC) Head Injury Study Group. CATCH: a clinical decision rule for the use of computed tomography in children with minor head injury. CMAJ. 2010 Mar 9;182(4):341-8. doi: 10.1503/cmaj.091421. Epub 2010 Feb 8. PMID 20142371
- [Background] Rogers AJ, Maher CO, Schunk JE, Quayle K, Jacobs E, Lichenstein R, Powell E, Miskin M, Dayan P, Holmes JF, Kuppermann N; Pediatric Emergency Care Applied Research Network. Incidental findings in children with blunt head trauma evaluated with cranial CT scans. Pediatrics. 2013 Aug;132(2):e356-63. doi: 10.1542/peds.2013-0299. Epub 2013 Jul 22. PMID 23878053
- [Background] Pearce MS, Salotti JA, Little MP, McHugh K, Lee C, Kim KP, Howe NL, Ronckers CM, Rajaraman P, Sir Craft AW, Parker L, Berrington de Gonzalez A. Radiation exposure from CT scans in childhood and subsequent risk of leukaemia and brain tumours: a retrospective cohort study. Lancet. 2012 Aug 4;380(9840):499-505. doi: 10.1016/S0140-6736(12)60815-0. Epub 2012 Jun 7. PMID 22681860
- [Background] Greenes DS, Schutzman SA. Clinical indicators of intracranial injury in head-injured infants. Pediatrics. 1999 Oct;104(4 Pt 1):861-7. doi: 10.1542/peds.104.4.861. PMID 10506226
- [Background] Palchak MJ, Holmes JF, Vance CW, Gelber RE, Schauer BA, Harrison MJ, Willis-Shore J, Wootton-Gorges SL, Derlet RW, Kuppermann N. A decision rule for identifying children at low risk for brain injuries after blunt head trauma. Ann Emerg Med. 2003 Oct;42(4):492-506. doi: 10.1067/s0196-0644(03)00425-6. PMID 14520320
- [Background] Jehlé E, Honnart D, Grasleguen C, et al. Comité de pilotage. Minor head injury (Glasgow Coma Score 13 to 15): triage, assessment, investigation and early management of minor head injury in infants, children and adults. Ann Fr Med Urg 2012;2:199-214